CLINICAL TRIAL: NCT02218177
Title: Neovascular Age-related Macular Degeneration: Intraocular Inflammatory Cytokines in the Non-responder to Ranibizumab Treatment
Brief Title: Intraocular Cytokines in Non-responders to Ranibizumab Treatment for Neovascular AMD
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Wai-Ching Lam, Professor University of Toronto, Residency Program Director Dept. of Ophthalmology, Continuing Medical Education Director Dept. of Ophthalmology, University Health Network, Toronto
Other Study IDs: VEGF wAMD cytokine study
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Age Related Macular Degeneration
Keywords: wet Age Related Macular Degeneration; Ranibizumab; Aflibercept; Combination Photodynamic Therapy; Cytokine analysis
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept; Ranibizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aqueous Humour from Eye
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-responders receiving aflibercept therapy: Non-responders to ranibizumab who are now receiving aflibercept therapy
  Interventions: Drug: Aflibercept
- Non-responders receiving PDT combo therapy: patients who are non-responders to ranibizumab who have been switched to combination photodynamic therapy (PDT)
  Interventions: Procedure: Combination Photodynamic Therapy
- Responders to ranibizumab: Patients who are responders to ranibizumab and are continuing monthly injections.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Aflibercept — anti-VEGF treatment for wet age related macular degeneration
  Other Names: Eylea (R)
  Groups: Non-responders receiving aflibercept therapy
Drug: Ranibizumab — anti-VEGF treatment for wet age related macular degeneration
  Other Names: Lucentis
  Groups: Responders to ranibizumab
Procedure: Combination Photodynamic Therapy — Use of cold laser with an intravitreal injection of dexamethasone to treat wet age related macular degeneration
  Groups: Non-responders receiving PDT combo therapy

SUMMARY:
The purpose of this study is to evaluate the level of cytokines (which are small proteins important in cell signalling) in eye fluid (aqueous humour) in patients with wet age related macular degeneration patients who have been treated with an injection in the eye (intravitreal injection) with a drug called ranibizumab. The level of cytokines will be compared between patients who have a good response to ranibizumab treatment and patients who are non-responsive to ranibizumab and need other forms of therapy. This knowledge will help for the future treatment and to potentially develop new medication for wet age-related macular degeneration.

DETAILED DESCRIPTION:
In the treatment of CNV (Choroidal NeoVascularization) secondary from AMD (Age Related Macular Degeneration) by using ranibizumab, patients who are non-responders can be found in approximately 1-10% of treatments. Thus, failure of treatment can lead to loss of vision. Growth factors and cytokines, such as vascular endothelial growth factor (VEGF), pigment epithelium derived factor (PEDF), interleukin 6 (IL-6) and placenta growth factor (PLGF) are known to play an important role in the development of CNV angiogenesis.

The rationale for conducting this study to compare VEGF, PEDF, IL-6 and PLGF cytokine levels in the aqueous humor of wet AMD and Polypoidal Choroidal Vasculopathy (PCV) patients who are poor responders to anti VEGF treatment and age-matched "good" responders to anti VEGF. Ranibizumab poor responders in AMD and PCV, who are treated with a combination of PDT/ranibizumab or intravitreous injection of aflibercept (Eyelea®, Regeneron Pharmaceuticals Inc. Tarrytown, NY, USA and Bayer, Basel, Switzerland) will be enrolled to the study. An aqueous humor sample will be obtained when patient receives intravitreal injection treatment and also at 1, 2 months follow up period. VEGF, PEDF,IL-6 and PLGF in aqueous will be analyzed and used to compare between the poor response group and age matched patient with good response to ranibizumab. Age, gender, visual acuity, central macular thickness by OCT, lesion size and fundus autofluorescence data will be collected and used to compare between these groups. Subgroup analysis of different treatment comparison with ranibizumab good responder group will be evaluated. Factors associated with the non-responders of ranibizumab will be analyzed.

Non-responders to ranibizumab treatment in AMD may have different levels and responses of inflammatory cytokines compared to the responder group. Understanding the pathogenesis and characteristic of this specific group of patients can help narrow down a specific choice of treatment and prevent the reduction of visual acuity of the patient. This study also helps identify factors associated to poor responders from ranibizumab treatment for wAMD.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or more
* Ranibizumab resistance/poor responder patients in all AMD entities (typical AMD, PCV and RAP) who will be treated with intravitreous ranibizumab in combination with verteporfin photodynamic therapy
* Ranibizumab resistance/poor responder patients in all AMD entity (typical AMD, PCV and RAP) who will be treated with intravitreous aflibercept injection
* AMD patient who is good response to the treatment of ranibizumab (control group)

Exclusion Criteria:

* Any evidence of good response in treatment of ranibizumab,
* Uncooperative patients to intravitreal treatment
* Patients who have clinically active ocular inflammation
* Patients who have previous PDT treatment within 6 months
* Patient who previously have ocular treatment of immunosuppressive agent within 3 months
* Patient who previously have ocular treatment of steroid with in 3 months
* Patients who are currently on systemic treatment of anti-VEGF medication or immunosuppressive agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study patients in the treatment group will be those greater than 50 years old, with age related macular degeneration, who are non-responder/ resistance to ranibizumab treatment. Control group will include patients who are responders to ranibizumab treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Aqueous Humour Cytokine Levels | At time of Intravitreal Injection

SECONDARY OUTCOMES:
Demographic Data | At time of appointment
Number of anti-VEGF injections before developing non-responder characteristics | At time of appointment
History of Previous Treatment | At time of appointment
Optical Coherence Tomography (OCT) results | At time of appointment
Fluorescein Angiography Results and Indocyanine Green Angiography Results | At time of appointment

CONTACTS AND LOCATIONS:
Overall Officials: Wai-Ching Lam, MD, Principal Investigator — Toronto Western Hospital, University Health Network, University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Pongsachareonnont P, Mak MYK, Hurst CP, Lam WC. Neovascular age-related macular degeneration: intraocular inflammatory cytokines in the poor responder to ranibizumab treatment. Clin Ophthalmol. 2018 Sep 26;12:1877-1885. doi: 10.2147/OPTH.S171636. eCollection 2018. PMID 30310267